CLINICAL TRIAL: NCT05668754
Title: A Phase 2, Placebo-Controlled, Double-Blind, Randomized Withdrawal Study to Determine the Safety and Efficacy of Oral SDX in Patients With Idiopathic Hypersomnia (IH)
Brief Title: Placebo-Controlled, Double-Blind, Study to Determine the Safety and Efficacy of SDX in Patients With IH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zevra Therapeutics (Industry)
Collaborators: Rho, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KP1077.D01
Record Dates: First submitted 2022-12-19; First posted 2022-12-30 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Idiopathic Hypersomnia
Keywords: Disorders of Excessive Somnolence; Sleep Disorders; Intrinsic Dyssomnias; Sleep Wake Disorders; Nervous System Diseases; Mental Disorders
MeSH Terms: conditions — Idiopathic Hypersomnia; Disorders of Excessive Somnolence; Sleep Wake Disorders; Nervous System Diseases; Mental Disorders | interventions — serdexmethylphenidate and dexmethylphenidate

STUDY DESIGN:
Intervention Model Description: Phase 2, placebo-controlled, double-blind, randomized withdrawal study to determine the safety and efficacy of oral SDX in patients with Idiopathic Hypersomnia (IH).
Who Masked: Participant, Investigator
Masking Description: Open-Label Titration Period with a Double-Blind Withdrawal Period
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Experimental: SDX (Experimental): SDX capsules at the optimized daily dose, once in the evening daily (qd pm) or twice per day (bid), for 2 weeks (DBWP)
  Interventions: Drug: Serdexmethylphenidate
- Active Comparator (Placebo Comparator): Placebo capsules once in the evening daily (qd pm) or twice per day (bid), for 2 weeks (DBWP)
  Interventions: Drug: Serdexmethylphenidate; Other: Placebo

INTERVENTIONS:
Drug: Serdexmethylphenidate — Participants randomized to active drug will receive their optimized dose according to a dosing regimen set by randomization at the start of the OLTP. The 4 possible oral SDX doses are 80, 160, 240, or 320 mg/day. The optimal SDX dose will be determined during the 5-week OLTP preceding the 2-week DBWP.
  Other Names: SDX
Other: Placebo — Participants randomized to placebo will receive matching placebo capsules to the optimized dose established at the end of the OLTP, according to a dosing regimen set by randomization at the start of the OLTP.
  Arms: Active Comparator

SUMMARY:
This is a study of the safety, efficacy and pharmacokinetics (PK) of Serdexmethylphenidate (SDX) compared to placebo in subjects with Idiopathic Hypersomnia (IH).

DETAILED DESCRIPTION:
SDX is a prodrug of dexmethylphenidate (d-MPH). SDX behaves as a prototypical prodrug that is devoid of pharmacological effects until metabolized to active d-MPH. Central nervous system (CNS) stimulants, including d-MPH products, are being used off-label by patients with IH. The potential advantage of SDX-derived d-MPH is its unique PK profile with rising d-MPH plasma concentrations at approximately 3 hours postdose followed by a broad peak from approximately 8 to 12 hours postdose (without sharp exposure spikes), and a gradual decline after the peak.

The optimal dose of SDX will be determined for each participant by titration based on individual tolerability and response during the 5-week SDX-only Open-Label Titration period (OLTP), after which 2/3 of the participants will continue to receive SDX and 1/3 of the participants will receive placebo (withdrawal design) in the 2-week Double-Blind Withdrawal Period (DBWP).

The study will evaluate safety (primary endpoint), efficacy and PK in patients with IH after daily oral administration of SDX either once per day in the evening (qd pm) or twice per day (morning and evening: bid). The study is expected to inform about the optimal SDX dose range and the best dose regimen (nighttime dosing or twice-per-day) for further studies in patients with IH and narcolepsy. The evening dosing regimen (just before bedtime) is of interest since there is little or no exposure to d-MPH for the first several hours post-dose and the mean peak d-MPH concentration occurs at 10-12 hours post-dose (ie, in the morning after a nighttime dose).

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age at the time of consent
2. Body Mass Index (BMI) ≤35 kg/m2
3. Documented primary diagnosis of IH according to the International Classification of Sleep Disorders (ICSD-3) criteria
4. At the Screening Visit and Baseline Visit (start of OLTP), Epworth Sleepiness Scale (ESS) scores ≥11
5. Average nightly Total Sleep Time (TST) of ≥7 hours, per subject history and confirmed during screening.
6. Subject must be in general good health defined as the absence of any clinically relevant abnormalities as determined by the Investigator based on physical and neurological examinations, vital signs, ECGs, medical history, and clinical laboratory values (hematology, chemistry, and urinalysis) at Screening.
7. If currently treated with nicotine replacement therapy, must have been taking the same regimen and dose for at least 2 months prior to screening and must agree to take the same dose during the study.
8. Have used a medically acceptable method of contraception for at least 2 months prior to the first dose of study drug and consent to use a medically acceptable method of contraception from the first dose of study drug, throughout the entire study period, and for 90 days after the last dose of study drug.

Exclusion Criteria

1. Hypersomnia due to another medical, behavioral, or psychiatric disorder condition (eg, narcolepsy, depression disorders, multiple sclerosis, Parkinson's disease, stroke).
2. Clinically significant sleep-related breathing disorders, including sleep apnea, treatment with Continuous Positive Airway Pressure (CPAP) therapy, Obstructive Apnea Hypopnea Index (AHI) >15 episodes per hour, or hypoventilation.
3. Clinically significant parasomnias (eg, sleep walking, rapid eye movement [REM] sleep behavior disorder, etc).
4. Periodic Limb Movement Disorder (PLMD) Arousal Index (PLMA-I) >15 during Screening PSG, a historical diagnosis of PLMD (last 10 years), or a PLMD diagnosis older than 10 years with current (last 60 days) treatment or symptoms of rhythmic movements involving one or both legs during sleep.
5. Occupation requiring nighttime shift work or variable shift work with early work start times (before 6 AM), if this occurs more than once per week.
6. Planned travel during the study that includes more than 3 time zones, or planned travel that includes 3 time zones on more than 2 occasions during the study.
7. Going to sleep for the night later than 1 AM at a frequency of more than once per week.
8. Current or past (within 1 year) major depressive episode according to DSM-5 criteria.
9. Any history of attempted suicide (lifetime) or clinically significant suicidal ideation, in the opinion of the Investigator, based on the C-SSRS assessment at Screening.
10. Any clinically significant unstable medical abnormality, chronic disease (eg, asthma or diabetes), or a history of a clinically significant abnormality of the cardiovascular, central nervous system,
11. Any of the following out-of-range vital signs at Screening: systolic blood pressure outside 90-145 mmHg; diastolic blood pressure outside 50-90 mmHg; resting heart rate outside 40-100 beats per minute.
12. History or presence of abnormal ECGs, which in the Investigator's opinion is clinically significant, including the following:

    1. ECG findings of ischemia or infarct
    2. Complete bundle branch blocks
    3. Symptomatic arrhythmias as ventricular arrhythmias (non- sustained ventricular tachycardia (VT), multifocal or frequent premature ventricular contractions), bundle branch block, axis deviation, or abnormal or any predominantly non-sinus- conducted rhythm.
    4. QTcF >450 msec for males or >470 msec for females, on Screening ECG.
    5. PR interval outside the range of 120 to 220 msec on Screening ECG
13. Estimated glomerular filtration rate (GFR) at Screening <60 mL/min/1.73 m2.
14. Malignant neoplastic disease requiring therapy within 2 years prior to Screening or during the study, or clinically relevant as judged by the Investigator.
15. Uncontrolled thyroid disorder as evidenced by thyroid stimulating hormone (TSH) ≤0.8 x the lower limit of normal (LLN) or ≥1.25 x the upper limit of normal (ULN) for the reference laboratory at Screening.
16. Laboratory value for aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 x upper limits of normal (ULN).
17. Excessive caffeine use during the 10 days prior to first dose of study drug or anticipated excessive use defined as >600 mg/day of caffeine during the treatment periods of the study.
18. Treatment or planned treatment with prohibited medications (including medications that may affect daytime sleepiness and nighttime sleep) or unwilling to refrain from any prohibited medications. Treatment must have been discontinued 14 days or 5 half-lives, whichever is longer, prior to the first dose of study medication (and at least 30 days for sedating antidepressants; at least 14 days for CNS stimulants).
19. Current or past (within 12 months prior to Screening) substance use disorder (including alcohol and psychoactive cannabinoids) according to DSM-5 criteria; current or past history of substance abuse treatment (including alcohol), or unwilling to refrain from substance use (including alcohol) during the study.
20. Nicotine dependence that has an effect on sleep (eg, a subject who routinely awakens at night to smoke).
21. Evidence of substance or alcohol use or has a positive urine or breath alcohol or positive urine drug screen at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-12-28 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-03-21 (Actual)

PRIMARY OUTCOMES:
Safety parameters - TEAEs | Time Frame: Start of OLTP to end of DBWP (7 weeks)
  Type and frequency of Treatment-Emergent Adverse Events
Safety parameter - Heart Rate | Time Frame: Start of OLTP to end of DBWP (7 weeks)
  Change from baseline in heart rate (beats/minute).
Safety parameter - Blood Pressure | Time Frame: Start of OLTP to end of DBWP (7 weeks)
  Change from baseline in blood pressure (mmHg).
Safety parameter - Laboratory Tests | Time Frame: Start of OLTP to end of DBWP (7 weeks)
  Clinical significant change from baseline in clinical laboratory tests.
Safety parameter - ECG | Time Frame: Start of OLTP to end of DBWP (7 weeks)
  Clinical significant change from baseline in electrocardiogram (ECG).
Safety parameter - PSQI | Time Frame: Start of OLTP to end of DBWP (7 weeks)
  Change from baseline in Pittsburg Sleep Quality Index Question #6. Sleep quality score ranging from very good (0) to very bad (4).

SECONDARY OUTCOMES:
Change from baseline in Epworth Sleepiness Scale (ESS) score | Start to end of DBWP (2 weeks)
  Scores level of daytime sleepiness ranging from 0 to 24, with a higher score indicating worsened sleepiness
Change from baseline in Brain Fog score | Time Frame: Start to end of DBWP (2 weeks)
  Queries for frequency, severity, and symptoms of cognitive impairment in the last week.
Percentage of participants with increase (worsening) of 2 points or more from baseline in the Clinical Global Impression of Severity (CGI-S) | Start to end of DBWP (2 weeks)
  Clinician-reported level of illness.
Percentage of participants with increase (worsening) of 2 points or more baseline in the Patient Global Impression of Severity (PGI-S). | Start to end of DBWP (2 weeks)
  Patient-reported level of illness.
Change from baseline in Total Score of the Idiopathic Hypersomnia Severity Hypersomnia Scale (IHSS) | Start to end of DBWP (2 weeks)
  Patient-reported questionnaire assessing the severity of excessive sleepiness, prolonged sleep duration, cognitive impairment and sleep inertia. The total score ranges from 0 to 50, with higher scores indicating more severe symptoms.
Change from baseline in Modified Karolinska Sleepiness Scale in the morning and late afternoon. | Start to end of DBWP (2 weeks)
  Patient-reported at-the-moment sleepiness, ranging from 1 (extremely alert) to 10 (extremely sleepy, can't keep awake).
Change from baseline in Patient-Reported Outcomes Measurement Information System-29 (PROMIS-29) total scores for depression, fatigue, and social functioning. | Start to end of DBWP (2 weeks)
  Queries functioning and well-being in the last week.
Change from baseline in the Patient-Reported Wakefulness Questionnaire (ZOGIM-A) total scores. | Start to end of DBWP (2 weeks)
  Queries alertness over the course of the day.
Change from baseline in the Sleep Inertia Visual Analog Scale (SIVAS) score. | Start to end of DBWP (2 weeks)
  Patient-reported measure of the difficulty of waking up in the morning, ranging from 0 (very easy) to 100 (very difficult)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Drake, PhD, Principal Investigator — Investigator
Locations (41):
- United States (41):
  - Sleep Disorders Center Of Alabama, Birmingham, Alabama
  - Amr Daphne, Daphne, Alabama
  - Lakeview Clinical Research, Guntersville, Alabama
  - SOCAL Clinical Research, Huntington Beach, California
  - Stanford University, Redwood City, California
  - Sleep Medicine Specialists of California, San Ramon, California
  - SDS Clinical Trials, Inc, Santa Ana, California
  - Delta Waves, Inc., Colorado Springs, Colorado
  - Saint Francis Sleep Allergy and Lung Institute LLC, Clearwater, Florida
  - New Generation of Medical Trials, Hialeah, Florida
  - Angels Clinical Research, Miami, Florida
  - Ivetmar Medical Group, Miami, Florida
  - Somnology Research Associates, Miami, Florida
  - Clinical Trial Services, Corp, Miami, Florida
  - Pasadena Center for Medical Research, St. Petersburg, Florida
  - Clinical Site Partners, LLC - Winter Park, Winter Park, Florida
  - Global Research Associates, Atlanta, Georgia
  - Neurotrials Research, Inc, Atlanta, Georgia
  - Clinical Research Institute - Stockbridge, Stockbridge, Georgia
  - The University of Kansas Medical Center Research Institution Inc., Kansas City, Kansas
  - Mid-Atlantic Epilepsy and Sleep Center - Bethesda, Bethesda, Maryland
  - Neurocare, Inc., Newton, Massachusetts
  - Western Michigan University Homer Stryker Md School of Medicine, Kalamazoo, Michigan
  - Henry Ford Health - Columbus, Novi, Michigan
  - Clinical Neurophysiology Services PC, Sterling Heights, Michigan
  - University of Missouri School Of Medicine, Columbia, Missouri
  - Clayton Sleep Institute, Llc, St Louis, Missouri
  - Barrett Clinic, La Vista, Nebraska
  - Global Medical Institutes LLC- Princeton Medical Institute, Lawrence, New Jersey
  - Clinical Research of Gastonia (CRG), Gastonia, North Carolina
  - Intrepid Research, Cincinnati, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Brian Abaluck, LLC, Malvern, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University Of South Carolina (MUSC) - Institute Of Psychiatry (IOP), Charleston, South Carolina
  - Bogan Sleep Consultants, Columbia, South Carolina
  - Futuresearch Trials Of Neurology, Austin, Texas
  - Dfw Clinical Research Associates, Fort Worth, Texas
  - Houston Clinical Research Associates, Houston, Texas
  - Sleep Therapy & Research Center, San Antonio, Texas
  - TPMG Clinical Research - Williamsburg, Williamsburg, Virginia